CLINICAL TRIAL: NCT04912570
Title: Thrombus Aspiration in Heavy Thrombus Burden Acute ST-elevation Myocardial Infarction: TSUNAMI Trial
Brief Title: Thrombus Aspiration in Heavy Thrombus Burden Acute ST-elevation Myocardial Infarction
Acronym: TSUNAMI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: No catheters
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIG0502101
Record Dates: First submitted 2021-05-19; First posted 2021-06-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; ST Elevation Myocardial Infarction
Keywords: Coronary Artery Disease; Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Thrombus Aspiration (Experimental): Manual Thrombus aspiration in STEMI patients with Heavy thrombus burden (TIMI 0-1 or TB classification 4-5)
  Interventions: Procedure: Manual Thrombus Aspiration
- Standard PCI (Active Comparator): Conventional PCI according to the most recent guidelines in STEMI patients with no heavy thrombus burden (TIMI 0-1 or TB classification 4-5)
  Interventions: Procedure: Standard PCI

INTERVENTIONS:
Procedure: Manual Thrombus Aspiration — Manual thrombus aspiration using one of the FDA approved aspirators will be done.
  Other Names: Thrombus Aspiration
  Arms: Manual Thrombus Aspiration
Procedure: Standard PCI — Standard PCI according to the most recent guidelines
  Arms: Standard PCI

SUMMARY:
Recent guidelines for the management of ST-elevation myocardial infarction (STEMI) recommend against the routine use of thrombus aspiration (TA) during primary percutaneous coronary intervention (PPCI) (Class III indication). Yet, so far, there is limited data regarding its role STEMI patients with heavy thrombus burden (TB).

The aim of this trial is to evaluate the effects of manual TA and PCI in comparison to conventional PCI alone in a real-life clinical trial among heavy TB STEMI patients undergoing PPCI.

DETAILED DESCRIPTION:
Recent guidelines for the management of ST-elevation myocardial infarction (STEMI) recommend against the routine use of thrombus aspiration (TA) during primary percutaneous coronary intervention (PPCI) (Class III indication). Yet, so far, there is limited data regarding its role in STEMI patients with heavy thrombus burden (TB).

The aim of this trial is to evaluate the effects of manual TA and PCI in comparison to conventional PCI alone in a real-life clinical trial among heavy TB STEMI patients undergoing PPCI.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients with heavy thrombus burden as assessed by TIMI score of 0-1 or thrombus burden classification 4-5

Exclusion Criteria:

* STEMI patients with low thrombus burden (TIMI 2-3 or TB 0-3)
* History of hypersensitivity or allergy to any of the study drugs, as well as known or suspected contraindications to the study drugs.
* Symptomatic hypotension and/or an SBP < 100 mmHg at the time of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Angiographic results | immediately after procedure
  Successful revascularization assessed by TIMI flow
Angiographic results | immediately after procedure
  Successful revascularization assessed by myocardial blush.
Angiographic results | immediately after procedure
  Successful revascularization assessed by ST-segment resolution.
In-hospital Major adverse cerebrovascular and cardiovascular events (MACCE) | 10 days
  Incidence of any major adverse cerebrovascular and cardiovascular events which includes: death (either all-cause or cardiac), nonfatal myocardial infarction, stroke and revascularization (with optional additional specification of target vessel or lesion, i.e., if the revascularization occurred at the site of a previously identified diseased coronary vessel or atherosclerotic lesion, respectively)
Short term Major adverse cerebrovascular and cardiovascular events (MACCE) | 6 months
  Incidence of any major adverse cerebrovascular and cardiovascular events which includes: death (either all-cause or cardiac), nonfatal myocardial infarction, stroke and revascularization (with optional additional specification of target vessel or lesion, i.e., if the revascularization occurred at the site of a previously identified diseased coronary vessel or atherosclerotic lesion, respectively) in the period of 6 months after randomization.

SECONDARY OUTCOMES:
Incidence of any bleeding event (Safety outcomes) | 10 days
  Incidence of any bleeding event that may be encountered during the hospital stay after randomization. (Major or Minor)
In-Hospital Heart failure status | 10 days
  Incidence of any event of heart failure that may be encountered during the hospital stay after randomization.
Short term Hospitalization due to heart failure | 6 months
  Incidence of any event of heart failure that may be encountered during any other re-admission due to a "heart failure" diagnosis up to 6 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Badran, MD, Study Chair — Ain Shams University, Egypt; Mahmoud H Abdelnabi, MD, Principal Investigator — University of Alexandria - Egypt; Ahmed M El Amrawy, MD, Study Director — University of Alexandria - Egypt; Yasser Sadek, MD, Study Director — National Heart Institute, Egypt
Locations (4):
- Egypt (4):
  - Andalusia Hospitals, Alexandria
  - International Cardiac Center (ICC), Alexandria
  - Ain Shams University Hospitals, Cairo
  - National Heart Institute, Giza